CLINICAL TRIAL: NCT06262373
Title: Are Early Pregnancies Implanted Close to the Tubal Ostia at Increased Risk of Miscarriage? A Prospective Observational Study
Brief Title: Angular Pregnancy - Ultrasound Definition and Correlation With Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 221321
Record Dates: First submitted 2023-04-25; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Miscarriage in First Trimester
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultrasound based observational study

SUMMARY:
The aim of this study is to establish clinically meaningful ultrasound-based diagnostic criteria for AP. To this end, the investigators will prospectively collect clinical and ultrasound data from early intrauterine pregnancies and correlate this data with pregnancy outcomes (particularly with risk of miscarriage), to establish whether there are any diagnostic criteria that can be used to make the diagnosis, facilitate increased surveillance of at risk pregnancies and reassure those with normally located pregnancies. The collected data will be used to correlate incidence of angular pregnancy and clinical variables such as maternal age, uterine fibroids, assisted conception, multiple pregnancy, ethnicity, previous uterine and adnexal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Have capacity to understand the study and to provide signed and dated informed consent.
* Willing to comply with all study procedures and be available for the duration of the study including consenting to follow up of the pregnancy outcome by letter, phone or email according to individual preference.
* Age 16 years or over
* Mean gestational sac diameter (GSD) on ultrasound of 2-15mm inclusive
* GS implantation site within the upper half of the uterine cavity on 2D USS

Exclusion Criteria:

* Women with pregnancies of unknown location, ectopic pregnancies or larger GSD than specified in the inclusion criteria.
* Implantation site within the lower half of the endometrial cavity on 2D USS screening.
* Intention to terminate the pregnancy
* Women with unicornuate uteri or unicornuate uteri with rudimentary horns
* Women with uterine fibroids which distort the uterine cavity

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women who are attending for a scan in the early pregnancy unit, aged over 16 years.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Primary | 2 years
  To define "angular pregnancy" using ultrasound based criteria.

SECONDARY OUTCOMES:
Secondary | 2 years
  To prospectively validate the ultrasound measurements that could be used to define implantation site in early pregnancy
Secondary | 2 years
  To correlate these measurements with pregnancy outcome (miscarriage vs no miscarriage)

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data is available for reasonable requests including study protocol and anonymised data.